CLINICAL TRIAL: NCT05298982
Title: Long-term Evaluation of Disability and Quality of Life at 1,2 and 5 Years in Invasively Mechanically Ventilated Patients Who Received Early Activity and Mobilisation Compared to Standard Care.
Brief Title: The TEAM Long-Term Cohort Study (A Sub-study of TEAM(III))
Status: Enrolling by invitation | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Medical Research Institute of New Zealand (Other); National Health and Medical Research Council, Australia (Other); ANZICS Clinical Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: U1111-1195-3567-A9
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Critically Ill; Mechanical Ventilation; Long Term Outcome
Keywords: Early activity and mobilization; rehabilitation; intensive care; health status
MeSH Terms: conditions — Critical Illness; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention arm: TEAM protocol: Based on TEAM (III) protocol patients will be assessed daily by an ICU physiotherapist using the ICU Mobility Scale (IMS) to determine the dosage and type of active exercises the patient will receive, using the early activity and mobilisation protocol. This protocol is hierarchical, with the objective of each intervention session beginning with the highest level of activity possible for the longest time possible, which then steps down to lower levels of activity if the patient fatigues. The intervention will be administered on all days in which the patient is admitted to ICU during the index hospitalisation, censored at 28days after.
  Interventions: Behavioral: Early activity and Mobilisation Intervention
- Standard of Care arm: TEAM protocol: Based on TEAM (III) protocol the control group will receive standard care from physiotherapy staff not involved in delivering the intervention. We have previously established that standard care in Australia for a patient receiving prolonged IMV (control group intervention) frequently involves no active exercise out of bed.

INTERVENTIONS:
Behavioral: Early activity and Mobilisation Intervention — The early activity and mobilisation intervention is comprised of exercises based on a reproducible, physiological approach using both strength and functional activities
  Groups: Intervention arm: TEAM protocol

SUMMARY:
This study is a prospective cohort study to evaluate the long-term effects of early activity and mobilisation compared to standard care on disability, function and health status for patients at 1, 2 and 5 years after recruitment of patients randomised into the TEAM Phase III RCT (ClinicalTrials.gov NCT03133377). The primary outcome of the study will be the level of disability as measured by the World Health Organisation's Disability Schedule 2.0, 12 level (WHODAS) at 2 years after recruitment.

DETAILED DESCRIPTION:
Incomplete recovery following critical illness is a major public health problem in Australia.

Each year around 150,000 Australians are admitted to intensive care (ICU). These critically ill patients require substantial resources and invasive, expensive interventions. Approximately 10% die and many of the remaining patients who survive have delayed and compromised functional recovery. As many as 25% of the ICU survivors who were living at home prior to ICU are unable to return home due to impaired physical function. Globally, the quality of survival following an ICU admission has been identified as one of the largest health challenges for these patients. This study will address the quality of survival and long-term functional recovery for patients who require life support in ICU. These patients account for 62% of the total bed-days in Australian ICUs, with direct care costs of $2 billion per year. The long-term outcomes for these patients are very poor. In my Australian cohort study, 50% of patients who survived hospital had disability

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the TEAM Phase III RCT Protocol.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 380 critically ill adult Australian patients, who met all of the inclusion criteria and none of the exclusion criteria, as defined in the TEAM Phase III RCT and consent to follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Level of disability measured with the World Health Organisation's Disability Assessment Schedule (WHODAS) 2.0 | Assessed 2 years after recruitment
  level of disability as measured by the World Health Organisation's Disability Schedule 2.0, 2 level (WHODAS) at 2 years after recruitment.

SECONDARY OUTCOMES:
Time from randomisation until death | From date of randomisation until date of death from all cause, censored at 5 years
All-cause mortality | From date of randomisation to 1 year
All-cause mortality | From date of randomisation to 2 years
All-cause mortality | From date of randomisation to 5 years
Generic function and disability measured using World Health Organisation's Disability Assessment Schedule (WHODAS) | Assessed 1 year after recruitment
Generic function and disability measured using World Health Organisation's Disability Assessment Schedule (WHODAS) | Assessed 5 years after recruitment
Quality of life and health status measured using the European Quality of Life 5 Dimensions 5 Level (EQ5D-5L) | Assessed 1 year after recruitment
Quality of life and health status measured using the European Quality of Life 5 Dimensions 5 Level (EQ5D-5L) | Assessed 2 years after recruitment
Quality of life and health status measured using the European Quality of Life 5 Dimensions 5 Level (EQ5D-5L) | Assessed 5 years after recruitment
Independent activities of daily living measured with The Lawton Instrumental Activities of Daily Living Scale (IADL) | Assessed 1 year after recruitment
Independent activities of daily living measured with The Lawton Instrumental Activities of Daily Living Scale (IADL) | Assessed 2 years after recruitment
Independent activities of daily living measured with The Lawton Instrumental Activities of Daily Living Scale (IADL) | Assessed 5 years after recruitment
Cognitive function measured using Montreal Cognitive Assessment (MOCA-Blind) | Assessed 1 year after recruitment
Cognitive function measured using Montreal Cognitive Assessment (MOCA-Blind) | Assessed 2 years after recruitment
Cognitive function measured using Montreal Cognitive Assessment (MOCA-Blind) | Assessed 5 years after recruitment
Psychological function measured using Hospital Anxiety and Depression scale | Assessed 1 year after recruitment
Psychological function measured using Hospital Anxiety and Depression scale | Assessed 2 years after recruitment
Psychological function measured using Hospital Anxiety and Depression scale | Assessed 5 years after recruitment
Psychological function measured using Impact of Event Scale - Revised (IES-R) | Assessed 1 year after recruitment
Psychological function measured using Impact of Event Scale - Revised (IES-R) | Assessed 2 years after recruitment
Psychological function measured using Impact of Event Scale - Revised (IES-R) | Assessed 5 years after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Prof Carol Hodgson, Study Chair — ANZIC-RC
Locations (16):
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - John Hunter Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Mater Health, Brisbane, Queensland
  - Mater Private Hospital, Brisbane, Queensland
  - Caboolture Hospital, Caboolture, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Launceston General Hospital, Launceston, Tasmania
  - Geelong Hospital - Barwon Health, Geelong, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sunshine Hospital, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] TEAM Study Investigators; Hodgson C, Bellomo R, Berney S, Bailey M, Buhr H, Denehy L, Harrold M, Higgins A, Presneill J, Saxena M, Skinner E, Young P, Webb S. Early mobilization and recovery in mechanically ventilated patients in the ICU: a bi-national, multi-centre, prospective cohort study. Crit Care. 2015 Feb 26;19(1):81. doi: 10.1186/s13054-015-0765-4. PMID 25715872
- [Background] Iwashyna TJ. Survivorship will be the defining challenge of critical care in the 21st century. Ann Intern Med. 2010 Aug 3;153(3):204-5. doi: 10.7326/0003-4819-153-3-201008030-00013. No abstract available. PMID 20679565
- [Background] Iwashyna TJ, Netzer G. The burdens of survivorship: an approach to thinking about long-term outcomes after critical illness. Semin Respir Crit Care Med. 2012 Aug;33(4):327-38. doi: 10.1055/s-0032-1321982. Epub 2012 Aug 8. PMID 22875378
- [Background] Higgins AM, Pettila V, Harris AH, Bailey M, Lipman J, Seppelt IM, Webb SA. The critical care costs of the influenza A/H1N1 2009 pandemic in Australia and New Zealand. Anaesth Intensive Care. 2011 May;39(3):384-91. doi: 10.1177/0310057X1103900308. PMID 21675057
- See also: TEAM study website — https://www.teamtrial.org.au/